CLINICAL TRIAL: NCT05674058
Title: Function and Imaging Assessments for G1961E-associated Stargardt Disease: Outcome Measure Ranking as Basis for Interventional Trials
Brief Title: Function and Imaging Assessments for G1961E-associated Stargardt Disease
Acronym: FIRSTORBIT
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: FIRSTORBIT
Record Dates: First submitted 2022-12-21; First posted 2023-01-06 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Stargardt Disease; Stargardt Disease 1; Fundus Flavimaculatus; Macular Degeneration, Stargardt; Macular Dystrophy With Flecks, Type 1
Keywords: Stargardt Disease; STGD1; p.Gly1961Glu; G1961E; c.5882G>A
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — According to clinical practice.

SUMMARY:
Some phenotypes of Stargardt disease are rather distinct. This includes the 'bull's eye maculopathy' phenotype associated with the frequent ABCA4 G1961E variant. In anticipation of a treatment trial, this natural history study aims to compare functional and structural outcome measures systematically.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with G1961E-associated Stargardt disease
* Defined by (1.) the presence of two pathogenic ABCA4 variants with at least one ABCA4G1961E variant, (2.) a Stargardt disease phenotype, and (3.) the absence of pathogenic variants in PRPH2, PROM1, and ELOVL4

Exclusion Criteria:

* Inability to give informed consent
* Prior surgery (other than anti-VEGF injections, cataract surgery, YAG laser capsulotomy, or laser retinopexy) that - according to the investigator's judgment - may affect visual function assessments (e.g., retinal detachment surgery, glaucoma filtration surgery, or a history of a corneal transplant in the study-eye)
* Concurrent ophthalmic conditions in the study eye that (according to the investigator's judgment) may contribute to loss of vision such as clinically significant opacification of the ocular media (corneal dystrophies, cataract), other retinal diseases, or disease of the optic nerve head and visual pathway (including amblyopia)
* Major surgery planned or other events that (according to the investigator's judgment) could hinder follow-up examinations (e.g., knee replacement)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include subjects with G1961E-associated Stargardt disease.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression of photoreceptor outer and inner segment loss | Two years from Baseline
  Rate of change for the (square-root transformed) EZ loss area (in mm/yr)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pfau M, Cukras CA, Huryn LA, Zein WM, Ullah E, Boyle MP, Turriff A, Chen MA, Hinduja AS, Siebel HE, Hufnagel RB, Jeffrey BG, Brooks BP. Photoreceptor degeneration in ABCA4-associated retinopathy and its genetic correlates. JCI Insight. 2022 Jan 25;7(2):e155373. doi: 10.1172/jci.insight.155373. PMID 35076026
- [Background] Pfau M, Holz FG, Muller PL. Retinal light sensitivity as outcome measure in recessive Stargardt disease. Br J Ophthalmol. 2021 Feb;105(2):258-264. doi: 10.1136/bjophthalmol-2020-316201. Epub 2020 Apr 28. PMID 32345606
- [Result] Maximilian Pfau, Georg Ansari, Giacomo Calzetti, Lucas Janeschitz-Kriegl, Bence Gyorgy, Kristina Pfau, Helene Dollfus, Carlo Rivolta, Hendrik PN Scholl; Fully Automated Patient-Tailored Microperimetry: FirstOrbit-Study Report. Invest. Ophthalmol. Vis. Sci. 2024;65(7):5403.